CLINICAL TRIAL: NCT03393559
Title: The Effect of Leg Elevation on the Prevention of Intraoperative Hypotension During Shoulder Surgery in the Beach Chair Position
Brief Title: Effect of Leg Elevation on Prevention of Intraoperative Hypotension During Beach Chair Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-1712-023-903
Record Dates: First submitted 2017-12-26; First posted 2018-01-08 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Intraoperative Hypotension; Cerebral Ischemia; Shoulder Disease
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Experimental): leg elevation during the beach chair position
  Interventions: Procedure: leg elevation
- Group C (No Intervention): Patients' leg will be straightened without any intervention.

INTERVENTIONS:
Procedure: leg elevation — Patients' leg will be raised by a pillow under both legs and the hip and knee joints will be flexed 45 degrees to position both knees at the heart level.
  Arms: Group L

SUMMARY:
The aim of this study is to evaluate the effect of leg elevation on the prevention of intraoperative hypotension during shoulder surgery in the Beach-chair position. patients undergoing shoulder surgery in the Beach-chair position will be randomly assigned to Group L (with leg elevation) or Group C (no intervention). The primary outcome is the incidence of intraoperative hypotension (mean blood pressure < 60mmHg or systolic blood pressure < 80% of baseline). Secondary outcomes are the incidence of intraoperative cerebral desaturation (cerebral oxygen saturation < 80% of baseline, longer than 30 seconds), total amounts of administered inotropic agents, and systolic blood pressure, heart rate, and cerebral oxygen saturation at various time points.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing shoulder surgery in the beach chair position

Exclusion Criteria:

* Patients with myocardial infarction
* Patients with pacemaker
* Patients with cerebrovascular disease
* patients with arteriovenous fistula at the opposite arm
* Patients with autonomic nerve disorders
* Patients with hip or knee joint disorder limiting hip or knee flexion
* BMI > 30 kg/m2

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative hypotension | From beach chair positioning to the end of surgery (average of 1 hour up to 2 hours)
  Mean blood pressure < 60 mmHg or systolic blood pressure < 80% of baseline

SECONDARY OUTCOMES:
Incidence of intraoperative cerebral desaturation | From beach chair positioning to the end of surgery (average of 1 hour up to 2 hours)
  Cerebral oxygen saturation < 80% of baseline longer than 30 seconds
Total amounts of administered inotropic agents | From beach chair positioning to the end of surgery (average of 1 hour up to 2 hours)
  Total amounts of administered inotropic agents after the Beach-chair positioning
Systolic blood pressure | before induction(baseline) / before the Beach-chair positioning / 1,5,30 and 60 minutes after the Beach-chair positioning
  Systolic blood pressure in mmHg at multiple time-points
Heart rate | before induction(baseline) / before the Beach-chair positioning / 1,5,30 and 60 minutes after the Beach-chair positioning
  Heart rate in bpm at multiple time-points
Peripheral oxygen saturation | before induction(baseline) / before the Beach-chair positioning / 1,5,30 and 60 minutes after the Beach-chair positioning
  Peripheral oxygen saturation in percentage at multiple time-points
Cerebral oxygen saturation | before induction(baseline) / before the Beach-chair positioning / 1,5,30 and 60 minutes after the Beach-chair positioning
  Cerebral oxygen saturation in percentage at multiple time-points

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available after article publication, for 3 years from the study completion.
Access Criteria: Proposals should be directed to the corresponding author and will be reviewed by the study group. Only requests that have a methodologically sound proposal and whose proposed use of the data has been approved by the independent review committee will be considered.

REFERENCES:
- [Derived] Nam S, Yoo S, Kim SH, Park SK, Lim YJ, Kim JT. Limited effect of leg elevation in preventing intraoperative hypotension during total shoulder arthroplasty in the beach chair position: a randomized controlled trial. BMC Anesthesiol. 2025 Oct 1;25(1):472. doi: 10.1186/s12871-025-03299-1. PMID 41034767